CLINICAL TRIAL: NCT03061916
Title: Antimicrobial Effects of Aqueous Extracts of Cinnamon and Ginger in Comparison to Chlorhexidine Gluconate 0.2% on Oral Streptococcus Mutans
Brief Title: Cinnamon and Ginger in Comparison to Chlorhexidine Gluconate 0.2% on Oral Streptococcus Mutans
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadhel Ahmed Mukred Mohamed, Master candidate at Conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: oper 606
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — ginger extract; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cinnamon (Experimental): 20% cinnamon will be given after collection of saliva (baseline) and samples will be taken after 30 minutes , one hour and two hours of giving cinnamon 20%
  Interventions: Dietary Supplement: Cinnamon
- Ginger (Experimental): 20% ginger will be given after collection of saliva (baseline) and samples will be taken after 30 minutes , one hour and two hours of giving ginger 20%
  Interventions: Dietary Supplement: Ginger
- Chlorhexidine (Active Comparator): Chlorhexidine gluconate 0.2%,will be given after collection of saliva (baseline) and samples will be taken after 30 minutes , one hour and two hours of giving chlorhexidine.
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Dietary Supplement: Cinnamon — Cinnamon 20% will be given to participants after baseline collection of saliva
  Other Names: Cinnamomum zeylanicum
  Arms: Cinnamon
Dietary Supplement: Ginger — Ginger 20% will be given to participants after baseline collection of saliva
  Other Names: Z. officinale
  Arms: Ginger
Drug: Chlorhexidine Gluconate — Chlorhexidine Gluconate will be given to participants after baseline collection of saliva
  Arms: Chlorhexidine

SUMMARY:
Chlorhexidine is the most potent chemotherapeutic agent against mutans streptococci and dental caries, however, the incidence of side effects such as teeth discoloration, staining of restorations, undesirable taste, discoloration of tongue, dryness and burning sensation in the mouth discourage patients to use this mouth wash. Natural products are now preferred by a large proportion of the population and have been reported to possess antimicrobial activity.These products have recently been shown to be a good alternative to synthetic chemical substances for caries prevention like Cinnamon and Ginger. The aim of this study is to compare the antimicrobial effects of aqueous extracts of cinnamon 20% and ginger 20% in comparison to chlorhexidine gluconate 0.2% on oral streptococcus mutans

DETAILED DESCRIPTION:
Sample Size Calculation The aim of this study is to compare the antimicrobial effects of aqueous extracts of cinnamon 20% and ginger 20% in comparison to chlorhexidine gluconate 0.2% on oral streptococcus mutans. 2 way with repeated measures analysis of variance will be performed to study the effect of different solutions at different times. Based on previous papers, a large effect size is expected (f=0.4). a minimum total sample size of 18 patients ( 6 in each group) will be sufficient with the power of 85% and a significance level of 5%. This number is to be increased to 21 to compensate for losses during follow up. The sample size was calculated using G*Power program (University of Dusseldorf, Dusseldorf, Germany). Recruitment Patient will be recruited from the outpatient clinic in the conservative department after explaining the benefits from the application of the interventions to their oral hygiene which is natural unlike other chemicals mouth rinses that has complications such as staining, and burning sensation; from which eligible patients will be recruited to fulfill the eligibility criteria.

Randomization:

Sequence generation:

Randomization will be computer generated using (www.randomization.com).

Allocation concealment:

Allocation of rinsing agents to groups will be done through sealed black opaque envelopes to ensure complete concealment.

Implementation:

A third party will perform the allocation sequence and assign the participants to rinsing agent in sequentially numbered opaque envelops.

Blinding:

The allocation group will be blinded from those assessing the outcome, data collectors, and data analysts. The microbiologists will be blinded by labeling the specimens with non-identifying terms.

Data collection methods:

Baseline data collection:

N.M will collect the baseline data through a chart which is composed of medical, dental history and clinical examination for every patient will be filled. The report will be anonymous where patients identified by their serial numbers (the first letter of the first and last name and date of birth) only will be registered. N.M will write the full detailed personal data of the patient in a separate sheet having the patient's serial number for further contact with patient, this sheet can only be seen by N.M. and the M.M.

Outcome data collection:

A microbiological technician will assess the viability counts of Mutans Streptococci in patients saliva at baseline and after 30 minutes, one hour and tow hours of rinsing.

Patient retention:

N.M. should understand the participant the final result will be expected and how it will differ in his/her oral hygiene. N.M. will told the participant that the whole procedure will take a short time and it will be painless.

Data management:

Data entry will be carried out by N.M. and revised by M.M.. All data will stored on computer and will be encrypted using a password. This will be done to allow accurate data entry through revision and protect data from being incorrectly used. Data will be packed up on another storage device to prevent it from being lost.

Statistical analysis :

Data will be analyzed using SPSS advanced statistics (Statistical Package for Social Sciences, version 21 (SPSS Inc. Chicago. IL). Numerical data will be described as mean and standard deviation or median and range. while qualitative data will be described as number and percentage. 2 way with repeated measures analysis of variance (ANOVA) will be performed. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

Data monitoring:

H.H. will monitor this study. Her role is to monitor any risk of bias could be done from participants, operator or assessors. Also to monitor blinding of the assessors and patient safety, outstanding benefits or harms.

Harms:

N.M. should inform participants about the possible harms, if present. Participants are allowed to contact the operator at moment through telephone. The data will be reported to N.M.

Auditing:

In the present trial, auditing will be done by the main and co-supervisors (H.H and M.M) to assure quality of the research methods and interventions. Ethics and dissemination

Research ethics approval:

Application forms for carrying out the clinical trial, checklist and informed consent of Research Ethics Committee (CREC) Faculty of Oral and Dental Medicine, Cairo University will be retrieved and filled, then will be delivered for (CREC) committee for approval, this is done to prevent any ethical problems during the study or any harm for any of the participants.

Protocol amendments:

If a new protocol will be used a protocol amendment will be submitted; containing a new copy of the new protocol and brief explanation about the differences between it and the previous protocols. If there is a change in the existing protocol that affect safety of subjects, investigation scope or scientific quality of the trial, an amendment containing a brief explanation about the change will be submitted. If a new author will be added to accomplish the study, an amendment including the investigator's data and qualifications to conduct the investigation will be submitted to prevent ghost authorship.

Consent or assent:

N.M. is responsible for admitting and signing the informed consents during the enrollment day.

Confidentiality:

Name and personal data of the participants will not appear on the protocol form and will be maintained secured for 10 years after the trial. This is done for protection of participants' privacy and civil rights.

Declaration of interests:

There is no conflict of interest, no funding or material supplying from any parties.

Access to data:

Access to final data will be allowed to the operator N.M. and main and co-supervisors (H.H. and M.M.) of the study who are involved in assessment of the outcome.

Ancillary and post-trial care:

Patients will not be followed up after intervention as there is no harm from our material we used .

Dissemination policy:

Full protocol will be published online in clinical trials website to avoid repetition and to keep the integrity of the research work. Thesis will be discussed in front of judgment committee. The study will be published to report the results of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Normal adults will be recruited in this study, all the volunteers participated in this experiment will be healthy looking with free medical history. The volunteers will be asked to suspend their usual oral hygiene practice at the day of the experiment

Exclusion Criteria:

* Volunteers that receives any antimicrobial agents during the last two weeks prior to study , wearing any fixed or removable prosthesis or orthodontic appliance will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-05-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
viability count measurement | within two hours
  The number of colonies will be expressed as colony-forming units multiplied by the dilution factor per milliliter of saliva (CFU/ml) and compared before and after rinsing

CONTACTS AND LOCATIONS:
Overall Officials: Heba Hamza, PhD, Study Director — Cairo university, Professor of conservative dentistry; Mai Mamdouh, PhD, Study Chair — Cairo university, lecturer of conservative dentistry
Locations (1):
- Nadhel Ahmed Mukred Mohamed, Cairo Governorate, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Azizi A, Aghayan S, Zaker S, Shakeri M, Entezari N, Lawaf S. In Vitro Effect of Zingiber officinale Extract on Growth of Streptococcus mutans and Streptococcus sanguinis. Int J Dent. 2015;2015:489842. doi: 10.1155/2015/489842. Epub 2015 Aug 12. PMID 26347778
- [Result] Hasan S, Danishuddin M, Khan AU. Inhibitory effect of zingiber officinale towards Streptococcus mutans virulence and caries development: in vitro and in vivo studies. BMC Microbiol. 2015 Jan 16;15(1):1. doi: 10.1186/s12866-014-0320-5. PMID 25591663
- [Result] Weli, Tuqa Akram, and Ahlam Taha Mohammed. Effect of ginger extract on Mutans streptococci in comparison to chlorhexidine gluconate. Journal of Baghdad College of Dentistry 25.2 (2013): 179-184.
- [Result] Al-Duboni, Ghada, Muhamed T. Osman, and R. Al-Naggar. Antimicrobial activity of aqueous extracts of cinnamon and ginger on two oral pathogens causing dental caries. Research Journal of Pharmaceutical, Biological and Chemical Sciences 4 (2013): 957-965.
- [Result] Rashad, J. M. Effect of water cinnamon extract on mutans streptococci, in comparison to chlorhexidine gluconate and zac (in vitro and in vivo study). Mustansiria Dent J 5 (2008): 250-60.